CLINICAL TRIAL: NCT00878631
Title: The Toronto Prehospital Hypertonic Resuscitation Head Injury and Multi Organ Dysfunction Trial
Brief Title: Feasibility Trial of Traumatic Brain Injured Patients Randomized in the Prehospital Setting to Either Hypertonic Saline and Dextran Versus Normal Saline
Acronym: TOPHR HIT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Sunnybrook Health Sciences Center, Toronto (Unknown); Defence Research and Development Canada (Industry)
Responsible Party: Laurie Morrison, St Michael's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TOPHR HIT; No.w7711-027801/001/TOR
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Last update posted 2009-04-09 (Estimated); Status verified 2009-04

CONDITIONS: Brain Injuries
Keywords: emergency medical services; traumatic brain injury; hypertonic saline with dextran; fluid resuscitation
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic | interventions — Dextrans; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Normal Saline (Active Comparator): infusion of 250 ccs of Normal Saline within 4 hours of the accident
  Interventions: Drug: Normal Saline
- 2 - hypertonic saline mixed with dextran (Experimental): a single dose 250 ml of 7.5% hypertonic saline in 6% dextran 70 infused within 4 hours of the accident
  Interventions: Drug: hypertonic saline mixed with dextran

INTERVENTIONS:
Drug: hypertonic saline mixed with dextran — a single dose 250 ml of 7.5% hypertonic saline in 6% dextran 70 is given within 4 hours from the time of the accident
  Other Names: RescueFlow BioPhausia AB, Stockholm Sweden
  Arms: 2 - hypertonic saline mixed with dextran
Drug: Normal Saline — 250 ccs of normal saline infused within 4 hours of the accident
  Arms: 1 Normal Saline

SUMMARY:
This clinical trial will evaluate the ease of conducting a randomized trial on patients with severe head injury who are cared for by paramedics in the out of hospital setting. The trial will compare two different kinds of fluids that are commonly used to elevate blood pressure and minimize the impact of the brain injury. The two solutions are a salt solution of different concentrations. One is a normal saline solution similar to the consistency of human blood and the other is a higher concentration mixed with a sugar that helps to keep the solution in the blood stream longer. This study is conducted without patient consent at the time of the study enrolment. The study will report on whether this trial is feasible in the out of hospital setting before launching into a larger definitive trial.

DETAILED DESCRIPTION:
The Toronto Prehospital Hypertonic Resuscitation-Head Injury and Multi Organ Dysfunction Trial (TOPHR HIT) is a randomized, placebo-controlled out of hospital trial of blunt trauma patients with head injuries. The study compares a group receiving normal saline according to a paramedic's protocol, with a treatment group receiving a single dose 250 ml of 7.5% hypertonic saline in 6% dextran 70 (RescueFlow BioPhausia AB, Stockholm Sweden).

The primary objective of this study is to report feasibility in accordance with the methodology described by Lancaster and Dodds*, specifically addressing:

1. baseline survival rates for the treatment and control group to aid in the design of a definitive multicentre trial.
2. randomization compliance rate.
3. ease of protocol implementation in the out-of-hospital setting.
4. adverse rate of HSD infusion.

The secondary objectives include measuring the effect of HSD in modulating the immuno-inflammatory response to severe head injury and its effect on modulating the release of neuro-biomarkers into serum; evaluating the role of serum neuro-biomarkers in predicting patient outcome and clinical response to HSD intervention; evaluating effects of HSD on brain atrophy post-injury and neurocognitive and neuropsychological outcomes.

*Lancaster, G.A., S. Dodd, and P.R. Williamson, Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract, 2004. 10(2): p. 307-12.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 16;
* Initial assessment of GCS 8 or less;
* Blunt traumatic mechanism of injury.

Exclusion Criteria:

* Known pregnancy;
* Primary injury penetrating;
* VSA prior to randomization;
* Previous Intravenous therapy ≥ 50 ml;
* Time interval between arrival at scene and intravenous access exceeds four hours;
* Amputation above wrist or ankle;
* Any burn (thermal, chemical, electrical, radiation)
* Suspected hypothermia;
* Asphyxia (strangulation, hanging, choking, suffocation, drowning)
* Fall from height ≤ 1m or ≤ 5 Stairs

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2004-09; Primary Completion 2006-01 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
baseline survival rates for the treatment and control group to aid in the design of a definitive multicentre trial | survival at 48 hours, hospital discharge, 30 days and 4 months
randomization compliance rate | duration of enrolment
ease of protocol implementation in the out-of-hospital setting | duration of study
adverse event rate of hypertonic saline dextran infusion | duration of study

SECONDARY OUTCOMES:
neurocognitive outcomes at discharge (cerebral performance category) and at 4 months (functional independence measure, disability rating scale, Glasgow Outcome Scale and Glasgow outcome Scale Extended | discharge and at 4 months post incident
neuropsychological outcomes including learning and memory, working memory, executive function, language function, visuospatial function, speed of processing and Beck Depression Scale. A focused attention reaction time test was added to 12 month testing. | at 4 and 12 months post incident
magnetic resonance imaging to evaluate effects of HSD on brain atrophy post-injury | 4 months post incident
the effect of HSD in modulating the immuno-inflammatory response to severe head injury and its effect on modulation the release of neuro-biomarkers into serum; evaluating the role of serum neuro-biomarkers in predicting patient outcome | samples taken within 48 hours of incident

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - St Michael's Hospital, Toronto, Ontario

REFERENCES:
- [Result] Morrison LJ, Rizoli S, Schwartz B, Rhind S, Black S, Stuss DT, Baker A, Univ of Toronto, Sunnybrook Health Sciences Centre, Toronto, Canada; on behalf of the TOPHR HIT Investigators. The Toronto Prehospital Resuscitation Head Injury and Multi-Organ Dysfunction Trial (TOPHR HIT). Circulation October 31, 2006; 114(18): #104.
- [Result] Morrison LJ, Rizoli S, Schwartz B, Rhind S, Black S, Stuss DT, Baker A, Stuss DT, Baker A, Simitciu M, Perreira T, MacDonald RD. University of Toronto, Sunnybrook Health Sciences Center, Toronto, Canada; on behalf of the TOPHR HIT Investigators. The Toronto Prehospital Hypertonic Resuscitation Head Injury and Multi-Organ Dysfunction Trial (TOPHR HIT). Prehosp Emerg Care 2007; 11(1): 94.
- [Derived] Rhind SG, Crnko NT, Baker AJ, Morrison LJ, Shek PN, Scarpelini S, Rizoli SB. Prehospital resuscitation with hypertonic saline-dextran modulates inflammatory, coagulation and endothelial activation marker profiles in severe traumatic brain injured patients. J Neuroinflammation. 2010 Jan 18;7:5. doi: 10.1186/1742-2094-7-5. PMID 20082712
- [Derived] Morrison LJ, Rizoli SB, Schwartz B, Rhind SG, Simitciu M, Perreira T, Macdonald R, Trompeo A, Stuss DT, Black SE, Kiss A, Baker AJ. The Toronto prehospital hypertonic resuscitation-head injury and multi organ dysfunction trial (TOPHR HIT)--methods and data collection tools. Trials. 2009 Nov 20;10:105. doi: 10.1186/1745-6215-10-105. PMID 19930566